CLINICAL TRIAL: NCT01595763
Title: Orientación Diagnóstica de la Trombosis Venosa Profunda en la Atención Primaria. Estudio de Coste Efectividad
Brief Title: Diagnostic Approach of Deep Vein Thrombosis in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TVP-2011-13
Record Dates: First submitted 2012-05-07; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Thrombosis
Keywords: Deep vein thrombosis; Primary care; Diagnosis; Clinical model
MeSH Terms: conditions — Thrombosis; Venous Thrombosis; Disease | interventions — fibrin fragment D; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood to calculate the value of Dimer D
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep Vein Thromobosis signs or symptoms
  Interventions: Other: D Dimer and ultrasonography

INTERVENTIONS:
Other: D Dimer and ultrasonography — clinical history, Dimer D, ultrasonography

SUMMARY:
To asses the cost-effectiveness of implementing different diagnostic strategies in patients with clinical assessment of suspected deep vein thrombosis (DVT) at first presentation in primary care. To evaluate the utility of using D dimer test to diagnose DVT in primary care. To describe the differential diagnosis and the strength of association between each outcome variable and the clinical prediction guide and the final diagnosis. It is a cross-sectional, multicentric study.

DETAILED DESCRIPTION:
The participants are the patients referred from the 15 primary care centers (400.000 inhabitants) to the Hospital de la Santa Creu i Sant Pau emergency department with suspected DVT. We will enter physical examination and anamnesis variables, Wells and Oudega's rules variables, D-Dimer value and ultrasonography result. The outcome variables are the cost (€) of each possible way of diagnostic approach and the effectiveness will be measured by the ultrasonography result, which confirms or excludes the diagnosis. The sample will include 437 patients. A decision tree will be developed to analyze the different diagnostic options in DVT cases, using standard notation.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by physicians with clinical suspicions of a first episode of deep vein thrombosis visited in emergency department of Hospital Santa Creu i Sant Pau

Exclusion Criteria:

* anticoagulant treatment
* patients who will not be able to follow control visit
* patients with oncologic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred by physicians with clinical suspicions of a first episode of deep vein thrombosis visited in emergency department of Hospital Santa Creu i Sant Pau
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-11

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Barcelona, Spain